CLINICAL TRIAL: NCT05471310
Title: Eye-tacking Method as a Diagnostic Tool for Assessment of Oculomotor Parameters (Gaze-holding Score, Scan Path, Visually Guided Saccades Etc) in Pediatric Patients With Ataxia Telangiectasia
Brief Title: Videoocular Assessment of Eye Movement Activity in an Ataxia Telangiectasia
Status: Completed | Type: Observational
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Other Study IDs: LB_03/17/22
Record Dates: First submitted 2022-04-07; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Ataxia Telangiectasia; Dysmetria
Keywords: Eye movements; Saccades; Unstable gaze holding; Rehabilitation
MeSH Terms: conditions — Ataxia Telangiectasia; Cerebellar Ataxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ataxia-telangiectasia (A-T) is a multisystem auto-somal recessive disorder linked to the A-T mutated gene (ATM) on chromosome 11q22-23, and characterized by progressive neural degeneration, immunodeficiency, and progressive ocular motor dysfunction. In previous studies, the quantitative description of the ocular motor deficits from clinical examination was limited to various defects in saccade and gaze control, dysmetric saccades, impairments of smooth pursuit, gaze holding, convergence, vestibular and optokinetic nystagmus slow phases, and cancellation of the vestibulo-ocular reflex. The aim of our research is to add existing findings with quantitative description of oculomotor patterns in A-T patients using videooculography (VOG).

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of ataxia telangiectasia,
* informed consent,
* stay at the Clinical Research Rehabilitation Center "Russkoe Pole" for 14 days.

Exclusion Criteria:

* epilepsy,
* poor visual acuity, inability to percept from a computer monitor,
* inability to hold head and posture satisfactory to perform the tasks,
* difficulty to obtain adequate recordings due to corrective lenses,
* visual field defects.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The young citizens of Russia suffered from ataxia telangiectasia.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Gaze holding task | baseline, during the intervention-rehabilitation course (once)
  A fixation task in which the subject will require to look at a target-a green circle (diameter ~1) sequentially presented at eccentric (15 rightward and leftward, 8 upward and downward) positions, each eccentric position being sustained for 20 s. Gaze-holding score will be assessed for each circle by approximating the gaze position coordinates by the least squares method to obtain the best correspondence using the fit function. The areas of the obtained ellipses, reflecting the spread of gaze position coordinates, will be determined for each of the four circle positions in each subject. Areas will be expressed in square visual degrees (sq. deg.)
Visual search task | baseline, during the intervention-rehabilitation course (once)
  Ten black circles (diameter ~1) will be presented on the monitor distributed pseudorandomly over the screen. Subjects will be instructed to count silently the number of points and give a verbal response. Study parameters: the performance time, the number of fixations, their durations, the total length of the scanning trajectory, and the saccade amplitude.
Visually guided saccade task | baseline, during the intervention-rehabilitation course (once)
  The subject will be required to follow a target jumping their gaze from one corner of the square to the next as quickly as possible as soon as a circle appeared; saccades will be required in order to do this (An image of a square with side length 10° will be presented on the monitor and a red circle (diameter ~1°) appeared in the corners sequentially in the clockwise direction.) Study parameters: the total number of saccades completed, the proportions of relatively accurate (A in the range 8.5-11.5°), hypometric (short, A < 8.5°), and hypermetric (long, A > 11.5°), and corrective saccades (occurring only after dysmetric saccades, 1.5° < A < 5°);

SECONDARY OUTCOMES:
Scale for the assessment and rating of ataxia | baseline, during the intervention-rehabilitation course (once)
  A clinical scale that is based on a semi-quantitative assessment of cerebellar ataxia on an impairment level.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander F. Karelin, PhD, Study Director — Clinical Rehabilitation Research Center "Russkoe pole"
Locations (1):
- Clinical Rehabilitation Research Center "Russkoe pole", Chekhov, Russia